CLINICAL TRIAL: NCT01629641
Title: Reliability and Validity of Goniometric iPhone Applications for the Assessment of Active Shoulder External Rotation
Brief Title: Reliability and Validity of Goniometric iPhone Applications
Status: Completed | Type: Observational
Sponsor: Texas Woman's University (Other)
Responsible Party: Sponsor
Other Study IDs: 17008
Record Dates: First submitted 2012-06-18; First posted 2012-06-27 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Shoulder Pain
Keywords: goniometry; outcome measures; shoulder assessment
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Normals: Texas Woman's University students from the School of Physical Therapy - Houston campus will be recruited to participate in this study. The participant will be excluded if they have pain in the shoulder on the day of testing, less than 90 degrees of active or passive shoulder abduction, less than 90 degrees of active or passive elbow flexion, have had any previous surgeries or procedures to either shoulder or identify by self-report any reason that they should not perform active external rotation at the shoulder.

SUMMARY:
The purpose of this study is to determine the test-retest and inter-rater reliability and concurrent validity of two iPhone goniometric applications in the measurement of active shoulder external rotation as compared to a standard manual goniometer. The scientific hypotheses for this study are as follows:

1. There will be significant Pearson correlations (>.8) to demonstrate test-retest reliability for each of the tools between the 1st and 2nd round of testing as assessed by novice testers.
2. There will be significant intra-class correlation coefficients (>.8) to demonstrate inter-rater reliability between the novice tester and the experienced tester for each of the three tools.
3. There will be significant Pearson correlations (>.8) to demonstrate concurrent validity between the standard goniometer and the photo capture application, the standard goniometer and the accelerometer-based application and the photo capture application with the accelerometer-based app. as assessed by novice testers.

DETAILED DESCRIPTION:
The purpose of this study is to determine the test-retest and inter-rater reliability and concurrent validity of two iPhone goniometric applications in the measurement of active shoulder external rotation as compared to a standard manual goniometer. This research is being done to determine if there are other more reliable, valid or innovative technological ways to measure active range of motion. Four testers (three entry-level doctoral students in physical therapy and one of two experienced physical therapists) will be measuring currently enrolled physical therapy doctoral students. The two experienced physical therapists are the principle investigator and the listed investigator who is a Physical Therapist. Two separate iPhone applications (DrGoniometer, which is based on photo capture and GetMyROM, which is based on the iPhone's internal accelerometer) and a standard manual goniometer will be used to measure the participants.

All potential participants will receive a cover letter describing the study via email. If the student is interested in participating they will report to the testing room (wearing a tank top (male or female) or asked to remove their top (male)) at one of the scheduled testing times. All testing will occur in a laboratory room on the TWU-Houston campus. The participant will be asked to review and sign an informed consent form. Any questions related to the study will be specifically asked at this time but may be asked at any time during the duration of the study. The primary investigator or any co-investigator will assign a confidential participant number to the participant at this time. Next the participant will be asked to complete a demographic form. If the participant answers "yes" to question 4, 5, 6 or 7, he/she will be eliminated from the study and asked not to participate. At this time, the participant will be randomly assigned to testing table 1, 2 or 3 (all three tables will follow the same basic procedure but the participant will be assessed by the table's assigned instrument first). Also, the side of testing (left or right) will be randomly selected. For example, a participant may be randomly assigned to table 1 (right shoulder). The participant will report to table 1, which is the iPhone DrGoniometer station...therefore they will be measured with this tool first. All of the testers (novice and expert) will be blinded to the outcomes of the other measures. Tester 1 (novice) will evaluate active right shoulder external rotation range of motion (ROM) with the iPhone DrGoniometer with a piece of tape covering the measurement reading. Tester 1 will then hand the iPhone to the blinded recorder, who will remove the tape, record the measurement, replace the tape and hand the iPhone back to Tester 1. Then the participant will be measured with GetMyROM (by novice 2) and then the standard goniometer (by novice 3) in random order. Tape will also be placed over the measurements on the iPhone for GetMyROM and the standard goniometer in the same manner that will be used with DrGoniometer. Next, the skilled tester will measure the participant with the instrument used at the assigned table. The participant will stay with this assigned table for the duration of the testing. Now the participant will be asked to stand up and move around before returning to the table for the 2nd round of testing. At least fifteen minutes from initial testing, the three initial novice testers will repeat their measurements in the previous order. All measurements and time of testing for the first measurement will be recorded by blinded investigators (recorders) and entered into a password protected computer and password protected Excel file which will only be known to the primary investigator. The file and computer will be locked in the primary investigator's office when data collection is not actively taking place. The data linking the participant number with the participant's name will only be known by the primary investigator and the recording investigators. The iPhones will not be linked to the internet during the testing and all images will be deleted after the data is recorded. The data will be recorded on to an Excel data printout. After each data collection session, the data will be entered into the file electronically.

Measurement of Shoulder External Rotation:

This study will follow a standard measurement testing procedure for assessing shoulder external rotation. The participant will be asked to wear either a tank-top (females or males) or no shirt (males). The participant will lie on their back on a padded plinth (table). The participant will asked to place their test shoulder in approximately 90 degrees of abduction (away from the body) and the elbow flexed (bent) to 90 degrees. The forearm is placed in neutral or midway between pronation/supination (long axis rotation) with approximately 2/3rds of the proximal the entire humerus is supported by the table. A towel will be placed under the humerus so the elbow is approximately at the level of the shoulder. In order to achieve this position, participants will be instructed via the following script:

1. Lie on your back on the plinth.
2. Move to the edge of the plinth towards me.
3. Let me position your arm and put a towel under it.
4. Bring your arm back towards the table, into external rotation, until you feel like you can't go any farther
5. Hold this position.

For the standard goniometer measurement, the axis of the goniometer will be placed on the center of the olecranon and the stationary arm of the goniometer will be perpendicular with the floor and the moving arm will bisect the ulna towards the ulnar styloid process. For DrGoniometer, a photo will be taken of the participant at the end of normal active ROM and the amount of range of motion will be calculated using the app. For GetMyROM, the iPhone will be placed perpendicular to the ground, as determined by the tester, and then the edge of the iPhone will be placed on the caudal border of the ulna. Expected normal range of motion is approximately 90 degrees of external rotation. The testers will be watching for movement substitutions: elbow extension (straightening), scapular elevation, tilting or protraction. If the tester notices any compensatory movement patterns, the participant will be asked to return to neutral and repeat the movement without compensation.

3 Three different iPhones will be used. These iPhones belong to the investigators. They will all be iPhone 4 version. All iPhone wireless and 3G connections will be disabled prior to data collection in order to reduce potential loss of confidentiality. All iPhones will use the same version of the applications and will not perform any updates to these applications. All iPhones will have the same version of software and will not update the software on the iPhone during the study. All iPhones will be password protected in order to reduce potential loss of confidentiality. At the end of each testing session, one of the PT investigators will assure that the photos have been deleted prior to reestablishing connectivity with the internet. In addition, all investigators signed a confidentiality statement.

ELIGIBILITY:
Inclusion Criteria:

* Current graduate student at Texas Woman's University. Must be enrolled in the DPT graduate program in Physical Therapy at the Houston campus.

Exclusion Criteria:

* The participant will be excluded if they have pain in the shoulder on the day of testing, less than 90 degrees of active or passive shoulder abduction, less than 90 degrees of active or passive elbow flexion, have had any previous surgeries or procedures to either shoulder or identify by self-report any reason that they should not perform active external rotation at the shoulder.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Texas Woman's University students from the School of Physical Therapy - Houston campus will be recruited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2012-01; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Active Shoulder External Rotation Range of Motion
  Range of Motion will be collected via two iPhone applications and a standard goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Katy Mitchell, PT, PhD, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's University, Houston, Texas, United States